CLINICAL TRIAL: NCT00832169
Title: An Open, Single Dose, Phase I Study of the Excretion of Radioactivity, Metabolism and Pharmacokinetics Following Oral Administration of [14C]AZD1386 to Healthy Male Volunteers
Brief Title: Investigation of Rate+Extent of Excretion of Radioactivity in Urine+Faeces After Oral Administration of [14C]AZD1386
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD, Medical Science Director, Emerging Analgesia, Neuroscience, AstraZeneca R&D Södertälje, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D5090C00015; EudractCT: 2008-006552-22
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Pain
Keywords: Pain
MeSH Terms: conditions — Pain | interventions — AZD1386

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD1386

INTERVENTIONS:
Drug: AZD1386 — 1 dose of oral solution

SUMMARY:
The aim of this study is to get information about absorption, distribution, metabolism and excretion as well as the tolerability and safety of AZD1386 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 18 - 30 and weight of 50 to 100 kilos.
* Healthy volunteer must have regular bowel movements (at least once daily)

Exclusion Criteria:

* History of psychiatric or somatic disease/condition, which may interfere with the objectives of the study as judged by the investigator.
* A family history of short QT syndrome or sudden cardiac death amongst first degree relatives.
* Any clinically important abnormalities in heart rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes.

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2009-01; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Excretion (rate+extent) of radioactivity in urine+faeces following oral administration of [14C]AZD1386 | Until >90% of predicted total radioactivity has been recovered
Pharmacokinetics of total radioactivity in plasma + unchanged AZD1386 in plasma Metabolite profile in plasma+excreta | Predose, + postdose 0.5h, 1h, 2h, 4h, 6h, 8h, 12h, 24h, 48h, 72h, 96h, 120h, 144hPredose + postdose 1h, 4h, 8h, 24h for excreta from predose (baseline) + postdose from 0h continously until 144h

SECONDARY OUTCOMES:
AZD1386 metabolites in plasma+excreta if feasable | Predose, 1h, 4h, 8h 24h
Safety + tolerability of AZD1386 | Predose, 2h, 6h, 12h, 24h, 48h, 168h

CONTACTS AND LOCATIONS:
Overall Officials: Raj Chetty, MD, Principal Investigator — AstraZeneca R&D, CPU Alderley Park, UK; Lars Ståhle, MD, Study Chair — AstraZeneca R&D, Södertälje, Sweden
Locations (1):
- Research Site, Macclesfield, CHESHIRE, United Kingdom